CLINICAL TRIAL: NCT07268118
Title: Randomized Control Trial for Pain Control With Topical Lidocaine for Cervical Ripening Balloon Placement
Brief Title: Pain Control for Cervical Ripening Balloon
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Little, Associate Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000734
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Labor Induction
Keywords: cervical ripening; cervical balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Topical lidocaine (Experimental)
  Interventions: Drug: topical vaginal application lidocaine gel
- Standard of care (No Intervention)

INTERVENTIONS:
Drug: topical vaginal application lidocaine gel — Application of topical vaginal lidocaine prior to cervical balloon ripening
  Arms: Topical lidocaine

SUMMARY:
No standard of care exists for pain management during cervical ripening balloon placement. The purpose of this study is to evaluate if vaginal topical lidocaine reduces pain related to cervical ripening balloon placement during induction of labor.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Gestational age ≥37 weeks
* Viable pregnancy
* Intact membranes
* English speaking
* Interested in cervical ripening balloon placement
* Able to provide consent

Exclusion Criteria:

* Allergy or sensitivity to lidocaine
* Patients that already have neuraxial anesthesia (i.e. spinal, epidural, combined spinal/epidural)
* Known uterine or cervical anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Patient-reported pain during cervical ripening balloon placement. | Within 24 hours of cervical balloon ripening
  Patient-reported pain score during cervical ripening balloon placement on a visual analog scale from 0 (no pain) to 10 (most pain).

IPD SHARING:
Plan to Share IPD: Undecided